CLINICAL TRIAL: NCT02484287
Title: Quality Control: A Prospective Analysis of External Ventricular Drain (EVD) Effectiveness
Brief Title: Quality Control: A Prospective Analysis of EVD Effectiveness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution prior to study completion
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 4890
Record Dates: First submitted 2015-06-23; First posted 2015-06-29 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Catheter Related Infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Integra External Drainage Catheter (Active Comparator): The Integra External Drainage Catheter non antibiotic-impregnated EVD catheter
  Interventions: Device: The Integra External Drainage Catheter.
- Ventriclear EVD Antibiotic Catheter (Active Comparator): The Ventriclear EVD Antibiotic Catheter antibiotic-impregnated EVD catheter
  Interventions: Device: The Ventriclear EVD Antibiotic Catheter
- Codman Bactiseal EVD Catheter Set (Active Comparator): The Codman Bactiseal EVD Catheter Set antibiotic-impregnated EVD catheter
  Interventions: Device: The Codman Bactiseal EVD Catheter Set

INTERVENTIONS:
Device: The Integra External Drainage Catheter. — Participants will be randomly assigned to receive 1 of 3 drains, to determine the efficacy of antibiotic-impregnated vs non antibiotic-impregnated EVD catheters, in the reduction of infection rates associated with EVD use.
  Arms: Integra External Drainage Catheter
Device: The Ventriclear EVD Antibiotic Catheter — Participants will be randomly assigned to receive 1 of 3 drains, to determine the efficacy of antibiotic-impregnated vs non antibiotic-impregnated EVD catheters, in the reduction of infection rates associated with EVD use.
  Arms: Ventriclear EVD Antibiotic Catheter
Device: The Codman Bactiseal EVD Catheter Set — Participants will be randomly assigned to receive 1 of 3 drains, to determine the efficacy of antibiotic-impregnated vs non antibiotic-impregnated EVD catheters, in the reduction of infection rates associated with EVD use.
  Arms: Codman Bactiseal EVD Catheter Set

SUMMARY:
The purpose and/or hypothesis: To decrease the amount of external ventricular drain (EVD) related catheter infections by comparing the efficacy of Oklahoma University Medicine standard EVD catheters, both impregnated and non-impregnated, in three principle areas: incidence of infection, cost analysis, and average durations of placement, all while maintaining the standards of technique.

DETAILED DESCRIPTION:
Experimental design: Track external ventricular drain (EVD) associated infections and through quality prospective analysis and compare the usage of standard catheters used by the department here at Oklahoma University, 1) the 35cm Codman Bactiseal rifampin and clindamycin impregnated catheter, 2) the Ventriclear EVD Antibiotic Catheter, and 3) the 36 cm Integra Hermatic large style ventricular catheter, in terms of incidence of infections, cost, duration of placement, and differences in placement technique.

Proposed procedure: Monitor for infections associated with and related to EVD placement in patients and assess if infections rates are affected by usage of antibiotic impregnated EVD catheters.

Importance of knowledge reasonably expected to result from the research: While use of sterile techniques and periprocedural antibiotics have traditionally been used to combat infection, infection rates remain above goal leading to the question of whether the antibiotic impregnated catheter should be added to the standard of care. With the knowledge gained, the investigators hope to decrease the amount of external ventricular drain related catheter infections and reduce use of prolonged antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require placement of external ventricular drain.

Exclusion Criteria:

* Prisoners and/or those who may be pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Cheema, MD, Principal Investigator — Associate Professor
Locations (1):
- Oklahoma University Medical Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Bohnstedt BN, Ziemba-Davis M, Edwards G, Brom J, Payner TD, Leipzig TJ, Scott JA, DeNardo AJ, Palmer E, Cohen-Gadol AA. Treatment and outcomes among 102 posterior inferior cerebellar artery aneurysms: a comparison of endovascular and microsurgical clip ligation. World Neurosurg. 2015 May;83(5):784-93. doi: 10.1016/j.wneu.2014.12.035. Epub 2014 Dec 23. PMID 25541085
- [Background] Lane B, Bohnstedt BN, Cohen-Gadol AA. A prospective comparative study of microscope-integrated intraoperative fluorescein and indocyanine videoangiography for clip ligation of complex cerebral aneurysms. J Neurosurg. 2015 Mar;122(3):618-26. doi: 10.3171/2014.10.JNS132766. Epub 2014 Dec 19. PMID 25526265
- [Background] Kulwin C, Bohnstedt BN, Payner TD, Leipzig TJ, Scott JA, DeNardo AJ, Cohen-Gadol AA. Aneurysmal acute subdural hemorrhage: prognostic factors associated with treatment. J Clin Neurosci. 2014 Aug;21(8):1333-6. doi: 10.1016/j.jocn.2013.12.010. Epub 2014 Jan 24. PMID 24679648
- [Background] Ziemba-Davis M, Bohnstedt BN, Payner TD, Leipzig TJ, Palmer E, Cohen-Gadol AA. Incidence, epidemiology, and treatment of aneurysmal subarachnoid hemorrhage in 12 midwest communities. J Stroke Cerebrovasc Dis. 2014 May-Jun;23(5):1073-82. doi: 10.1016/j.jstrokecerebrovasdis.2013.09.010. Epub 2013 Oct 19. PMID 24144595
- [Background] Cohen-Gadol AA, Bohnstedt BN. Recognition and evaluation of nontraumatic subarachnoid hemorrhage and ruptured cerebral aneurysm. Am Fam Physician. 2013 Oct 1;88(7):451-6. PMID 24134085
- [Background] Bohnstedt BN, Nguyen HS, Kulwin CG, Shoja MM, Helbig GM, Leipzig TJ, Payner TD, Cohen-Gadol AA. Outcomes for clip ligation and hematoma evacuation associated with 102 patients with ruptured middle cerebral artery aneurysms. World Neurosurg. 2013 Sep-Oct;80(3-4):335-41. doi: 10.1016/j.wneu.2012.03.008. Epub 2012 Mar 30. PMID 22465372

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ventriclear EVD Antibiotic Catheter | Integra External Drainage Catheter | Codman Bactiseal EVD Catheter Set
Started | 15 | 26 | 19
Completed | 0 | 0 | 0
Not Completed | 15 | 26 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ventriclear EVD Antibiotic Catheter | Integra External Drainage Catheter | Codman Bactiseal EVD Catheter Set | Total
Number analyzed (Participants) | 15 | 26 | 19 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 9 | 17 | 12 | 38
  >=65 years | 5 | 9 | 7 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 8 | 31
  Male | 5 | 13 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 4
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 8
  White | 10 | 21 | 12 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 15 | 26 | 19 | 60

OUTCOME MEASURES:

1. Primary Outcome: Infection Rates of EVD Patients
Description: Infection rates of EVD patients
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ventriclear EVD Antibiotic Catheter | Integra External Drainage Catheter | Codman Bactiseal EVD Catheter Set
Number analyzed (Participants) | 15 | 26 | 19
Participants | 0 | 0 | 0

2. Other Pre Specified Outcome: Duration of EVD Placement
Description: duration of EVD placement in days
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Integra External Drainage Catheter | Ventriclear EVD Antibiotic Catheter | Codman Bactiseal EVD Catheter Set
Number analyzed (Participants) | 26 | 15 | 19
days | 11 (7) | 13 (10) | 10 (5)

3. Other Pre Specified Outcome: Cost
Description: Comparable cost of each device
Time Frame: 24 months
Population: This data was not collected and is no longer available.
Arm/Group | Ventriclear EVD Antibiotic Catheter | Integra External Drainage Catheter | Codman Bactiseal EVD Catheter Set
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 90 days (admission to discharge)
Description: Adverse events, specifically infections due to EVD were collected while participant was in the hospital.
Arm/Group | Integra External Drainage Catheter | Ventriclear EVD Antibiotic Catheter | Codman Bactiseal EVD Catheter Set
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 0/26 | 0/15 | 0/19

LIMITATIONS AND CAVEATS:
Recruitment was halted prematurely, due to changes in key study personnel. PI left prior to completing final data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT02484287/Prot_SAP_000.pdf